CLINICAL TRIAL: NCT00928161
Title: Evaluation and Treatment of Reflux Disease in Patients With Head and Neck Cancer Undergoing Radiation Therapy That Causes Significant Mucositis in the Reflux Field and Xerostomia
Brief Title: Reflux Disease in Head and Neck Cancer Patients Undergoing Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0944
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer; Gastroesophageal Reflux Disease
Keywords: Reflux Disease; Acid-reflux; Head and Neck Cancer; HNC; Radiation Therapy; Mucositis; Radiation-induced xerostomia; RIX; Dry Mouth; Heartburn; Dexlansoprazole; Prevacid; Prevacid Solu-Tab; GERD
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Gastroesophageal Reflux; Mucositis; Xerostomia; Heartburn | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (No Intervention): Patients with no acid reflux.
- Group 2 (Active Comparator): Patients with acid reflux.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dissolving tablet taken by mouth (60 mg tablet), once a day. Take dose first thing in morning on empty stomach, then nothing but water for 30-45 minutes afterwards.
  Other Names: Prevacid; Prevacid Solu-Tab
  Arms: Group 2

SUMMARY:
The goal of this clinical research study is to learn if radiation-induced xerostomia [RIX] (dry mouth) causes, or worsens the effects of, acid reflux (heartburn and heartburn-like symptoms) in head and neck cancer (HNC) patients receiving radiation therapy.

Objectives:

Primary Objective:

Determine if radiation induced xerostomia (RIX) increases the frequency or duration of acid-reflux when re-measured approximately 6-12 weeks after RT (measured by # episodes, their duration, and Reflux Area Index (RAI). Reflux Area (RA) is the sum of the area under the curve for all episodes of pH<4 recorded during the study in units of Ph*minutes. The Reflux area index (RAI) is the RA corrected for the duration of the study (RA x 100/study duration).

Secondary Objectives:

1. To demonstrate that patients undergoing RT for OPC have reflux into the irradiated field that is anticipated to exacerbate mucositis symptoms
2. Correlate RAI and # episodes of acid reflux with salivary flow before and after RT to determine if radiation induced hyposalivation is associated with more reflux events and symptoms.
3. For patients with no pre-RT pathologic acid reflux, determine if RIX leads to conversion to acid-positive reflux measured approximately 6-12 weeks after RT.
4. Correlate office indirect laryngoscopy findings (posterior commissure thickening, cobble-stoning, granulomas, and arytenoids erythema or edema) suggestive of acid reflux in OPC patients with pH-probe findings as was done in larynx cancer (Lewin et al)
5. Compare findings from the patient reported outcome (PRO) instruments used

DETAILED DESCRIPTION:
The Study Drug:

Dexlansoprazole is designed to block the production of excess stomach acid that is the cause of acid reflux disease.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 groups, based on the results of your screening tests.

If you are assigned to Group 1, you will not receive any study drug, but you will complete the study visits and radiation therapy, as described below.

If you are assigned to Group 2, you will receive Dexlansoprazole.

Study Drug Administration:

Dexlansoprazole is an dissolving tablet that is taken by mouth. It dissolves on the tongue. It should not be swallowed whole with water like a regular pill. You will take 1 tablet, once daily. The study drug should be taken first thing in the morning on an empty stomach, and then you should not eat or drink anything but water for 30-45 minutes after taking the study drug.

Study Visits:

Before you have the scheduled radiation therapy, you will have study visits. At these visits, the following tests and procedures will be performed:

* You will have a pH-probe test performed.
* You will complete the PRO questionnaires.
* You will have a whole mouth salivary flow (WMSF) test. To perform this test, you will chew a piece of non-flavored gum, and spit into a cup for after about 5 minutes. The amount saliva will be weighed and recorded to compare it the amount recorded after radiation therapy.

Radiation Therapy:

After you have completed the study visits, you will have the scheduled radiation therapy. You will be asked to sign a separate consent form for this.

Length of Study:

You will remain on study from the beginning of radiation therapy until the 6-12 week follow up visit is completed. After your participation on this study is over, you should speak with your primary doctor about long term treatment. If your acid reflux disease gets worse while on study, you will be recommended for a gastrointestinal (GI) evaluation and treatment. If you experience intolerable side effects, you will be taken off study.

Follow-Up Visits:

About 6-12 weeks after you have completed radiation therapy, you will have a follow up visit. At this visit, the following tests and procedures will be performed:

* You will have a pH-probe test performed.
* You will complete the PRO questionnaires.

This is an investigational study. Dexlansoprazole is FDA approved and commercially available for the treatment of acid reflux disease.

Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Head and neck cancer (HNC) Oropharynx cancer (OPC) patients who are adults > 18 years of age, dispositioned to receive curative RT with bilateral neck (including) parotid irradiation with or without chemotherapy.
3. Radiation Therapy (3D conformal or IMRT).

Exclusion Criteria:

1. Subjects unable to tolerate pH-probe in past.
2. Subjects currently on proton-pump inhibitor (PPI), daily antacids and daily H2 antagonists.
3. Prior history of esophago-gastric surgery.
4. Symptoms of active gastrointestinal bleeding (melena, hematemesis).
5. Known hepatic cirrhosis or esophageal varices.
6. Prior esophageal perforation.
7. Pregnant or lactating woman. Women of childbearing potential who have not undergone a hysterectomy with either a positive or no pregnancy test at baseline. Women / men of childbearing potential not using a reliable and appropriate contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
8. Subjects with allergies or sensitivities to proton-pump inhibitors.
9. Patients who cannot complete study follow-up and compliance with study protocol.
10. Patients on Plavix (if medically appropriate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of acid reflux episode (during each 24 hour pH probe) | Before radiotherapy and again at 6 weeks following radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: David I. Rosenthal, MD, MA, BA, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org